CLINICAL TRIAL: NCT03388996
Title: The Role of Pelvic Microbiomes During the Malignant Transformation of Benign Ovarian Diseases
Brief Title: Pelvic Microbiomes of Benign and Malignant Ovarian Diseases
Acronym: MTBOD-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Collaborators: Academy Military Medical Science, China (Industry)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: MTBOD-1
Record Dates: First submitted 2017-12-22; First posted 2018-01-03 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Microbiota; Ovarian Neoplasms; Ribosome Alteration
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Microbiota

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Discharges/flushing fluid from vagina, faces and fimbria end of fallopian tube are going to sent for analysis of 16s RNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign ovarian disease: The group consists of patients of benign ovarian diseases and health conditions (eg infertility), who would accept the tests of pelvic microbiomes.
  Interventions: Diagnostic Test: microbiomes
- Malignant ovarian disease: The group consists of patients of high grade serous carcinoma, who would accept the tests of pelvic microbiomes.
  Interventions: Diagnostic Test: microbiomes

INTERVENTIONS:
Diagnostic Test: microbiomes — 16s RNA analysis and microculture of discharges/flushing fluid from vagina, faces and fimbria end of fallopian tube

SUMMARY:
This case-control study aims to compare the pelvic microbiomes of benign ovarian diseases and ovarian malignancies by 16s RNA techniques and culture. Discharges/flushing fluid from vagina, faces and fimbria end of fallopian tube are collected from age and menopausal status matched patient before and during procedures of laparoscopies. The discharges/flushing fluid would be sent for 16s RNA analysis and microculture respectively, and the results would get self-contrasted comparison and case-control comparison.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopy procedures
* Specific pathological diagnosis

Exclusion Criteria:

* Previous history of pelvic surgeries
* Evidences of pelvic inflammation diseases

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group of benign ovarian diseases: patients with definite benigh ovarian diseases or health conditions (eg infertlity)
  Group of malignant ovarian diseases: patients with definite diagnosis of high grade serous carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Difference of species distribution of microorganism according to 16s RNA analysis | 2 years
  The difference of species of microorganism distribution according to 16s RNA sequencing analysis between control group and study group, and between different sampling sites in each arm
Difference of species distribution of microorganism according to microculture outcomes | 2 years
  Difference of species distribution of microorganism according to microculture outcomes between control group and study group, and between different sampling sites in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We would share individual participant data to all other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For ever